CLINICAL TRIAL: NCT00135421
Title: A Multicenter, Randomized, Double-Blind, Placebo and Escitalopram Controlled Trial of the Safety and Efficacy of BMS-562086 in the Treatment of Outpatients With Major Depressive Disorder
Brief Title: Study of BMS-562086 in the Treatment of Outpatients With Major Depressive Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN148-007
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2008-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — pexacerfont; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1 (Experimental)
  Interventions: Drug: Pexacerfont
- A2 (Active Comparator)
  Interventions: Drug: Escitalopram
- A3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pexacerfont — Tablets & Capsules, Oral, 100 mg, Once daily, Up to 8 weeks followed by 8 weeks of observation
  Other Names: BMS-562086
  Arms: A1
Drug: Escitalopram — Tablets & Capsules, Oral, 20 mg, Once daily, Up to 8 weeks followed by 8 weeks of observation.
  Arms: A2
Drug: Placebo — Tablets & Capsules, Oral, 0 mg, Once daily, Up to 8 weeks followed by 8 weeks of observation.
  Arms: A3

SUMMARY:
The purpose of this clinical research study is to learn whether BMS-562086 is both safe and effective in treating outpatients with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient women meeting Diagnostic and Statistical Manual of Mental Disorders Manual, Fourth Edition, Text Revision (DSM-IV TR) criteria for a single or recurrent, non-psychotic episode of Major Depressive Disorder (296.2x and 296.3x).
* Patients whose current depressive episode is at least three months in duration at the Baseline Visit.

Exclusion Criteria:

* Males
* Patients with treatment resistance to other antidepressants

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2005-11; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to endpoint (Week 8) on the total score of the Hamilton Depression Rating Scale (HAMD-17) | Week 8

SECONDARY OUTCOMES:
Compare safety and tolerability of BMS-562086 to placebo by assessing adverse events, vital signs, electrocardiograms (ECGs), physical examinations and clinical lab tests | every visit and endpoint
Compare efficacy of escitalopram to placebo | at endpoint and at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (45):
- United States (45):
  - Apc Clinical Research Trials Nw, Pa, Springdale, Arkansas
  - Pacific Clinical Research Medical Group, Orange, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Front Range Clinical Research, Wheat Ridge, Colorado
  - University Of Connecticut Health Center, Farmington, Connecticut
  - University Of Florida, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Cunningham Clinical Research, Llc, Edwardsville, Illinois
  - Alexian Center For Psychiatric Research, Hoffman Estates, Illinois
  - American Medical Research, Inc., Oak Brook, Illinois
  - Alpine Clinic, Lafayette, Indiana
  - J. Gary Booker, Md, Shreveport, Louisiana
  - Dupont Clinical Research, Rockville, Maryland
  - Summit Research Network, Farmington Hills, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Albuquerque Neuroscience, Inc., Albuquerque, New Mexico
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Bioscience Research, Llc, New York, New York
  - Social Psychiatry Research Institute, New York, New York
  - Behavioral Medical Research Of Staten Island, Staten Island, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Richard H. Weisler, Md, Raleigh, North Carolina
  - Community Research, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Oregon Center For Clinical Investigations, Inc. (Occi, Inc), Portland, Oregon
  - Summit Research Network, Portland, Oregon
  - Suburban Research Associates, Media, Pennsylvania
  - Usc School Of Medicine, Columbia, South Carolina
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Futuresearch Trials, Austin, Texas
  - Claghorn-Lesem Research Clinic, Bellaire, Texas
  - Insite Clinical Research, DeSoto, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Croft, Harry A., San Antonio, Texas
  - Radiant Research, Salt Lake City, Salt Lake City, Utah
  - University Of Utah School Of Medicine, Salt Lake City, Utah
  - Psychiatric Alliance Of The Blue Ridge, Charlottesville, Virginia
  - Dominion Clinical Research, Midlothian, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Summit Research Network (Seattle), Inc., Seattle, Washington
  - Northbrooke Research Center, Brown Deer, Wisconsin
  - Dean Foundation For Health Research & Education, Middleton, Wisconsin